CLINICAL TRIAL: NCT00453505
Title: Modulation of Motor Function by Stimulation of the Central and Peripheral Nervous System
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 070122; 07-N-0122
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2025-06-11

CONDITIONS: Motor Function of Healthy Physiology
Keywords: Transcranial Direct Current Stimulation; Transcranial Magnetic Stimulation; Peripheral Nerve Stimulation; Primary Motor Cortex; Corticomotor Excitability; Healthy Volunteer; HV
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- 1 (Experimental): Healthy Volunteers
  Interventions: Device: TMS
- 1a (Sham Comparator): Healthy Volunteers
  Interventions: Device: TMS
- 2 (Experimental): Healthy Volunteers
  Interventions: Device: tDCS
- 2a (Sham Comparator): Healthy Volunteers
  Interventions: Device: tDCS
- 3 (Experimental): Healthy Volunteers
  Interventions: Device: tACS
- 3a (Sham Comparator): Healthy Volunteers
  Interventions: Device: tACS
- 4 (Experimental): Healthy Volunteers
  Interventions: Device: CPNS
- 4a (Sham Comparator): Healthy Volunteers
  Interventions: Device: CPNS

INTERVENTIONS:
Device: TMS — <=1 Hz TMS for up to 30mins and up to 115% of resting motor threshold intensity (MT).
  Arms: 1; 1a
Device: tDCS — tDCS up to 2 mA for up to 60mins.
  Arms: 2; 2a
Device: tACS — tACS up to 1 mA for up to 10 minutes.
  Arms: 3; 3a
Device: CPNS — CPNS alone with intensities below 130% of the peripherally-elicited-motor-threshold for up to 2 hours.
  Arms: 4; 4a

SUMMARY:
Objectives

Noninvasive stimulation of the central and peripheral nervous system, including transcranial magnetic stimulation (TMS), transcranial direct and alternating current stimulation (tDCS and tACS, respectively) and cutaneous/peripheral nerve stimulation (C/PNS) alone or paired with TMS (paired associative stimulation, PAS), has been increasingly used in the investigation of cortical plasticity and as a possible adjuvant strategy in neurorehabilitation. It has been shown that TMS, tDCS, tACS and C/PNS can modulate motor function in healthy volunteers, as well as in patients with neurological disorders such as stroke.

One fundamental problem is that the optimal parameters of stimulation to modulate motor function by all of these techniques are not known. The purpose of this protocol is to explore within safe guidelines, the effects of different stimulation parameters on motor cortical function, on oscillatory brain dynamics measured with magnetoencephalography (MEG) and electroencephalography (EEG), on eye movements, and on fMRI activation. In addition, this protocol will be used to train new fellows coming to NINDS Human Cortical Physiology Section (HCPS) in the use of TMS, tDCS, tACS and C/PNS techniques.

We expect that information emerging from these studies will allow us to 1) optimize experimental protocols or stimulation parameters to collect pilot data in healthy volunteer for future patient-oriented hypothesis-driven protocols,2)to collect pilot data for power analysis for future patient-oriented hypothesis driven protocols, and 3) to train new fellows in the use of these different methods.

Study Population

Up to 1500 healthy volunteers, age 18 and older.

Design

Healthy volunteers will receive one or more of the following types of stimulation alone or in combination: (1) single- and paired-pulse TMS with inter-stimulus intervals of greater than 1s and up to 20s and intensities of up to 100% of stimulator output; (2) 1 Hz TMS for up to 30mins and up to 115% of resting motor threshold (RMT) intensity; (3) tDCS applied at an intensity of up to 4 mA for a duration of up to 60mins, as long the total charge does not exceed 7.2 C; (4) tACS applied at a peak-to-peak intensity of up to 4 mA for a duration of up to 60 minutes, minutes, as long the total charge does not exceed 7.2 C; (5) C/PNS applied alone with intensities below 130% of the peripherally-elicited-motor-threshold for up to 2 hours, or intensities up to 300% of sensory threshold when C/PNS is paired with TMS. All of these parameters of stimulation and procedures have safely been used as previously reported in the literature. Sham stimulations will be delivered for each modality as scientifically needed. Some substudies may involve recording of behavior or brain activity only (such as behavioral testing, MRI, and MEG) if brain stimulation targets are unknown. This information can help design future brain stimulation protocols.

Each subject may participate in up to 20 sessions. A single session may last no longer than 8 hours to allow for initial testing paradigm followed by retests or performing other components of the same substudy later in the day. Appropriate rest breaks and meal breaks will occur during long sessions. Subjects participate in one experimental session per day under this protocol. The 20 experimental sessions will be scheduled over a twenty-year period. CTDB is used to track the number of sessions per subject so it does not exceed 20 sessions. The AIs are responsible for entering the subjects/sessions into CTDB.

We will test the effects of these different forms of stimulation on motor cortical excitability, cognitive and motor behavioral tasks, and brain state measures derived from neuroimaging data (i.e. - MRI, fMRI, MEG and EEG). Stimulation may be applied before, after, or during physiological (i.e. motor evoked potentials, M-wave, F-wave, or H-Reflexes), neuroimaging or behavioral measures.

Under this protocol, we conduct:

Exploratory Sub-studies: These substudies are exploratory in nature and are conducted in order to develop information to generate better informed future hypotheses and/or power analyses. We have set an upper limit of 40 subjects per sub-study.

Hypothesis-Testing Sub-studies: Hypothesis-testing sub-studies are studies with specific hypotheses to be tested. These sub-studies undergo statistical and PIRC review after 6 subjects per group (e.g., after 12 subjects, 6 per arm, if two groups are studied), before additional subjects can be recruited. Together, the P.I. and PIRC will decide whether to continue the sub-study with more subjects without an amendment or whether an amendment or protocol would be necessary. A memo requesting a review of hypothesis-testing sub-studies for possible additional enrollment (beyond 6) will be sent to PIRC and the statistical reviewer.

This protocol is ...

DETAILED DESCRIPTION:
Objectives

Noninvasive stimulation of the central and peripheral nervous system, including transcranial magnetic stimulation (TMS), transcranial direct and alternating current stimulation (tDCS and tACS, respectively) and cutaneous/peripheral nerve stimulation (C/PNS) alone or paired with TMS (paired associative stimulation, PAS), has been increasingly used in the investigation of cortical plasticity and as a possible adjuvant strategy in neurorehabilitation. It has been shown that TMS, tDCS, tACS and C/PNS can modulate motor function in healthy volunteers, as well as in patients with neurological disorders such as stroke.

One fundamental problem is that the optimal parameters of stimulation to modulate motor function by all of these techniques are not known. The purpose of this protocol has been to explore within safe guidelines, the effects of different stimulation parameters on motor cortical function, on oscillatory brain dynamics measured with magnetoencephalography (MEG) and electroencephalography (EEG), on eye movements, and on fMRI activation. In addition, this protocol was used to train new fellows coming to NINDS Human Cortical Physiology Section (HCPS) in the use of TMS, tDCS, tACS and C/PNS techniques.

We expected that information emerging from these studies would allow us to 1) optimize experimental protocols or stimulation parameters to collect pilot data in healthy volunteers for future patient-oriented hypothesis-driven protocols, 2) to collect pilot data for power analysis for future patient-oriented hypothesis driven protocols, and 3) to train new fellows in the use of these different methods.

As instructed, we had stopped recruitment under this protocol at the time we were informed by the NIH IRB that they determined this to be a thematic protocol (August 6, 2019). The four specific aims addressed under this protocol are:

1. Aim 1. To identify resting behavioral and physiological substrates for neuromodulation of motor behavior
2. Aim 2. To identify task-dependent behavioral and physiological substrates for neuromodulation of motor behavior
3. Aim 3. To understand variability, rigor or/and reproducibility of brain stimulation effects.

As instructed, the purpose of this amendment is to request authorization to proceed with data analysis and publication. No new experiments will be carried out under this protocol.

Study Population

Up to 1500 healthy volunteers, age 18 and older.

Design

No new experiments will be carried out under this protocol. Previously, healthy volunteers received one or more of the following types of stimulation alone or in combination: (1) single- and paired-pulse TMS with inter-stimulus intervals of greater than 1s and up to 20s and intensities of up to 100% of stimulator output; (2) 1 Hz TMS for up to 30mins and up to 115% of resting motor threshold (RMT) intensity; (3) tDCS applied at an intensity of up to 4 mA for a duration of up to 60mins, as long the total charge does not exceed 7.2 C; (4) tACS applied at a peak-to-peak intensity of up to 4 mA for a duration of up to 60 minutes, as long the total charge does not exceed 7.2 C; (5) C/PNS applied alone with intensities below 130% of the peripherally-elicited-motor-threshold for up to 2 hours, or intensities up to 300% of sensory threshold when C/PNS is paired with TMS. All of these parameters of stimulation and procedures have safely been used as previously reported in the literature. Sham stimulations were delivered for each modality as scientifically needed. Some sessions included recording of behavior or brain activity (such as behavioral testing, MRI, and MEG) if brain stimulation targets were unknown. This information was used to inform the design of brain stimulation protocols.

Each subject was able to participate in up to one experimental session per day, and up to 20 total sessions over a twenty year period under this protocol. A single session lasted no longer than 8 hours. Appropriate rest breaks and meal breaks occured during long sessions. CTDB was used to track the number of sessions per subject to ensure they did not exceed 20 sessions. Protocol AIs were responsible for entering the subjects/sessions into CTDB.

We previously tested the effects of different forms of stimulation on motor cortical excitability, cognitive and motor behavioral tasks, and brain state measures derived from neuroimaging data (i.e. - MRI, fMRI, MEG and EEG). Stimulation was be applied before, after, or during physiological (i.e. motor evoked potentials, M-wave, F-wave, or H-Reflexes), neuroimaging or behavioral measures.

Outcome Measures

No new outcome measures are proposed. Changes in motor cortical excitability were previously measured as the change in the average peak-to-peak amplitude of a motor evoked potential (MEP) as measured with EMG. Neuroimaging measures included changes in oscillatory brain activity power as measured with EEG or MEG, changes in BOLD fMRI activation or changes in functional connectivity (i.e. covarying fluctuations in BOLD or spectral power across the brain). Behavioral outcome measures focused on changes in performance as a function of learning, or as a function of applied brain stimulation.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 18 and older
  2. Willingness and ability to give consent
  3. Normal neurological examination
  4. Clearly dominant handedness (right or left) as assessed by Handedness scales

EXCLUSION CRITERIA:

1. Any severe or progressive neurological disorder or severe medical condition, or history of seizures
2. Chronic use of medications acting primarily on the central nervous system, which lower the seizure threshold or significantly alter cortical excitability such as antipsychotic drugs (chlorpromazine, clozapine), tricyclic or other antidepressants, or prescription stimulants.
3. Pacemakers or other implanted electrical devices, brain stimulators, some types of dental implants, aneurysm clips (metal clips on the wall of a large artery), metallic prostheses (including metal pins and rods, heart valves, and cochlear implants), permanent eyeliner, implanted delivery pump, or shrapnel fragments
4. Diagnosis of drug dependence made by a health care provider (ICD-9-CM code 304)
5. Staff from our section

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1007 (Actual)
Dates: Start 2007-01-14 (Actual); Primary Completion 2019-11-08 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
To identify task-dependent behavioral and physiological substrates for neuromodulation of motor behavior Aim | in data analysis
  in data analysis
To understand variability, rigor or/and reproducibility of brain stimulation effects. | in data analysis
  in data analysis
To identify resting behavioral and physiological substrates for neuromodulation of motor behavior Aim | in data analysis
  in data analysis

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo G Cohen, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wassermann EM. Risk and safety of repetitive transcranial magnetic stimulation: report and suggested guidelines from the International Workshop on the Safety of Repetitive Transcranial Magnetic Stimulation, June 5-7, 1996. Electroencephalogr Clin Neurophysiol. 1998 Jan;108(1):1-16. doi: 10.1016/s0168-5597(97)00096-8. PMID 9474057
- [Background] Pascual-Leone A, Valls-Sole J, Wassermann EM, Hallett M. Responses to rapid-rate transcranial magnetic stimulation of the human motor cortex. Brain. 1994 Aug;117 ( Pt 4):847-58. doi: 10.1093/brain/117.4.847. PMID 7922470
- [Background] Muellbacher W, Ziemann U, Boroojerdi B, Hallett M. Effects of low-frequency transcranial magnetic stimulation on motor excitability and basic motor behavior. Clin Neurophysiol. 2000 Jun;111(6):1002-7. doi: 10.1016/s1388-2457(00)00284-4. PMID 10825706
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-N-0122.html